CLINICAL TRIAL: NCT04752904
Title: Noninvasive Continuous Blood Pressure Monitoring for Preventing Post-spinal Hypotension During Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Noninvasive Continuous Blood Pressure Monitoring for Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sun-Kyung Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2010-093-1165
Record Dates: First submitted 2021-02-05; First posted 2021-02-12 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Cesarean Section Complications; Hypotension
Keywords: noninvasive continuous blood pressure monitoring
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: randomized double blind controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ClearSight group (Experimental): Non-invasive, continuous blood pressure is monitored using ClearSight Sytem, with a finger cuff around the middle finger, and the anesthesiologist manages blood pressure based on this.
  Interventions: Device: ClearSight System
- Control group (No Intervention): The blood pressure is measured at 1-minute intervals by non-invasive blood pressure monitor using the arm cuff, and the anesthesiologist in charge manages the blood pressure based on the measured blood pressure.

INTERVENTIONS:
Device: ClearSight System — Non-invasive, continuous blood pressure is monitored using ClearSight Sytem
  Arms: ClearSight group

SUMMARY:
Noninvasive continuous blood pressure monitoring for preventing post-spinal hypotension during cesarean delivery: A randomized controlled trial

DETAILED DESCRIPTION:
The aim of this study was to find out whether the incidence of hypotension during surgery can be reduced in the case of non-invasive, continuous blood pressure monitoring using the ClearSight System in patients undergoing cesarean section under spinal anesthesia, compared to the case of using conventional noninvasive blood pressure monitoring

ELIGIBILITY:
Inclusion Criteria:

* Adult mothers who are pregnant with single fetuses over 35 weeks gestational age undergoing planned cesarean delivery under spinal anesthesia

Exclusion Criteria:

* Multiple fetal pregnancy

  * Preexisting hypertension or pregnancy-induced hypertension

    * Underlying heart disease

      * Underlying cerebrovascular disease

        * Known fetal anomaly

          * Contraindicated in spinal anesthesia

            * Any sign of onset of labor

              * Body weight <45 kg or body weight> 90 kg

                * Height <145cm or height> 180cm

                  * All other cases in which researchers determine to be inappropriate for this clinical trial

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension by individualized methods | From spinal anesthesia to delivery
  Hypotension was defined as: SBP<80% of baseline SBP

SECONDARY OUTCOMES:
Incidence of hypotension by standard methods | From spinal anesthesia to delivery
  Hypotension was defined as MBP<65mmHg
Time-weighted average SBP<80% of baseline SBP | From spinal anesthesia to delivery
  Time-weighted average SBP<80% of baseline SBP
Time-weighted average MAP <65mmHg | From spinal anesthesia to delivery
  Time-weighted average MAP <65mmHg
Incidence of intraoperative severe hypotension | From spinal anesthesia to delivery
  Defined as: SBP < 70% of baseline SBP
Incidence of intraoperative symptomatic hypotension | From spinal anesthesia to delivery
  Defined as: hypotension plus nausea and/or vomiting and/or dizziness and/or breathlessness
Incidence of nausea, vomiting, dizziness, breathlessness | From spinal anesthesia to delivery
  Incidence of nausea, vomiting, dizziness, breathlessness
Incidence of intraoperative Hypertension | From spinal anesthesia to delivery
  SBP> 120% of baseline SBP
Maximum, Minimum recorded SBP, DBP, MBP | From spinal anesthesia to delivery
  Maximum, Minimum recorded SBP, DBP, MBP
Cumulative duration of hypotension | From spinal anesthesia to delivery
  Cumulative duration of hypotension
Number of hypotensive episodes | From spinal anesthesia to delivery
  Number of hypotensive episodes
Onset time of hypotension | From spinal anesthesia to delivery
  Onset time of hypotension
Cumulative consumptions of vasopressors | From spinal anesthesia to delivery
  Cumulative consumptions of vasopressors
Incidence of bradycardia | From spinal anesthesia to delivery
  HR (heart rate) <50 bpm
Incidence of atropine use | From spinal anesthesia to delivery
  Incidence of atropine use
Minimum heart rate | From spinal anesthesia to delivery
  Minimum heart rate
Cardiac output, stroke volume | From spinal anesthesia to delivery
  only in ClearSight System group
The analysis of the differences between the test method (ClearSight) and reference method | From spinal anesthesia to delivery
  Bland-Altman analysis
Apgar Score | at 1 minute after delivery and 5 minutes after delivery
  1 minute, 5 minutes
Umbilical arterial blood | within 10 minutes after delivery
  Arterial blood gas analysis results
Umbilical arterial pH | within 10 minutes after delivery
  <7.2

CONTACTS AND LOCATIONS:
Overall Officials: Sun-Kyung Park, M.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wei C, Qian J, Zhang Y, Chang X, Hu H, Xiao F. Norepinephrine for the prevention of spinal-induced hypotension during caesarean delivery under combined spinal-epidural anaesthesia: Randomised, double-blind, dose-finding study. Eur J Anaesthesiol. 2020 Apr;37(4):309-315. doi: 10.1097/EJA.0000000000001152. PMID 31977628
- [Background] Hasanin AM, Amin SM, Agiza NA, Elsayed MK, Refaat S, Hussein HA, Rouk TI, Alrahmany M, Elsayad ME, Elshafaei KA, Refaie A. Norepinephrine Infusion for Preventing Postspinal Anesthesia Hypotension during Cesarean Delivery: A Randomized Dose-finding Trial. Anesthesiology. 2019 Jan;130(1):55-62. doi: 10.1097/ALN.0000000000002483. PMID 30335625
- [Background] Fitzgerald JP, Fedoruk KA, Jadin SM, Carvalho B, Halpern SH. Prevention of hypotension after spinal anaesthesia for caesarean section: a systematic review and network meta-analysis of randomised controlled trials. Anaesthesia. 2020 Jan;75(1):109-121. doi: 10.1111/anae.14841. Epub 2019 Sep 18. PMID 31531852
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Juri T, Suehiro K, Kimura A, Mukai A, Tanaka K, Yamada T, Mori T, Nishikawa K. Impact of non-invasive continuous blood pressure monitoring on maternal hypotension during cesarean delivery: a randomized-controlled study. J Anesth. 2018 Dec;32(6):822-830. doi: 10.1007/s00540-018-2560-2. Epub 2018 Sep 28. PMID 30267340
- [Background] Bartels K, Esper SA, Thiele RH. Blood Pressure Monitoring for the Anesthesiologist: A Practical Review. Anesth Analg. 2016 Jun;122(6):1866-79. doi: 10.1213/ANE.0000000000001340. PMID 27195632
- [Background] Rogge DE, Nicklas JY, Schon G, Grothe O, Haas SA, Reuter DA, Saugel B. Continuous Noninvasive Arterial Pressure Monitoring in Obese Patients During Bariatric Surgery: An Evaluation of the Vascular Unloading Technique (Clearsight system). Anesth Analg. 2019 Mar;128(3):477-483. doi: 10.1213/ANE.0000000000003943. PMID 30649073
- [Background] Noto A, Sanfilippo F, De Salvo G, Crimi C, Benedetto F, Watson X, Cecconi M, David A. Noninvasive continuous arterial pressure monitoring with Clearsight during awake carotid endarterectomy: A prospective observational study. Eur J Anaesthesiol. 2019 Feb;36(2):144-152. doi: 10.1097/EJA.0000000000000938. PMID 30562226
- [Background] Ngan Kee WD, Lee SWY, Ng FF, Lee A. Norepinephrine or phenylephrine during spinal anaesthesia for Caesarean delivery: a randomised double-blind pragmatic non-inferiority study of neonatal outcome. Br J Anaesth. 2020 Oct;125(4):588-595. doi: 10.1016/j.bja.2020.05.057. Epub 2020 Jul 15. PMID 32682556
- [Background] Vos JJ, Poterman M, Mooyaart EA, Weening M, Struys MM, Scheeren TW, Kalmar AF. Comparison of continuous non-invasive finger arterial pressure monitoring with conventional intermittent automated arm arterial pressure measurement in patients under general anaesthesia. Br J Anaesth. 2014 Jul;113(1):67-74. doi: 10.1093/bja/aeu091. Epub 2014 Apr 15. PMID 24740992
- [Background] Lawicka M, Malek A, Antczak D, Wajlonis A, Owczuk R. Non-invasive haemodynamic measurements with Nexfin predict the risk of hypotension following spinal anaesthesia. Anaesthesiol Intensive Ther. 2015;47(4):303-8. doi: 10.5603/AIT.2015.0048. PMID 26401736
- [Background] Chen G, Chung E, Meng L, Alexander B, Vu T, Rinehart J, Cannesson M. Impact of non invasive and beat-to-beat arterial pressure monitoring on intraoperative hemodynamic management. J Clin Monit Comput. 2012 Apr;26(2):133-40. doi: 10.1007/s10877-012-9344-2. Epub 2012 Mar 1. PMID 22382920
- [Background] Juri T, Suehiro K, Kimura A, Mukai A, Tanaka K, Yamada T, Mori T, Nishikawa K. Impact of continuous non-invasive blood pressure monitoring on hemodynamic fluctuation during general anesthesia: a randomized controlled study. J Clin Monit Comput. 2018 Dec;32(6):1005-1013. doi: 10.1007/s10877-018-0125-4. Epub 2018 Mar 6. PMID 29511971